CLINICAL TRIAL: NCT06085677
Title: The Gastric HormonE BioMarkers of Preneoplastic Lesions (GEM) Study
Brief Title: The Gastric HormonE BioMarkers of Preneoplastic Lesions Study
Acronym: GEM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Collaborators: University College, London (Other); University of Oxford (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: 23IC8542
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Stomach Neoplasm; Chronic Atrophic Gastritis; Intestinal Metaplasia
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal/mild gastritis: Patients enrolled with normal stomach epithelium or mild gastritis
- Chronic atrophic gastritis: Patients enrolled with chronic atrophic gastritis
- Intestinal metaplasia: Patients enrolled with intestinal metaplasia

SUMMARY:
The goal of the study is to understand whether blood levels of hormones produced or metabolized in the stomach reflect the health of the stomach lining.

Specifically the study will determine whether the concentration of ghrelin, gastrin, pepsinogens and vitamin B12 reflect the condition of the stomach lining. Hormone concentrations for people with normal/mild gastritis will be compared to people with long-term inflammation of the stomach (chronic atrophic gastritis), and people with pre-cancerous cellular changes (intestinal metaplasia).

DETAILED DESCRIPTION:
Previously published promising data show that blood levels of ghrelin, gastrin, vitamin B12 and pepsinogen are each associated with risk of developing stomach cancer. These studies used blood bank samples and looked at risk of cancer many decades later. This study was designed to explore whether these markers could be useful in a clinical setting for early detection of stomach cancer.

The study will recruit at 3 sites over 1 year identifying patients with chronic atrophic gastritis and intestinal metaplasia and those with mild gastritis.

Only the patient data which is absolutely necessary for analysis will be collected, to include basic demographics, relevant medical history and medications. These data will be used to analytically account for alternative explanations for variation in blood measurements of ghrelin, gastrin, pepsinogen and vitamin B12.

A one-time venous blood sample will be collected to enable measurement of the markers of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-80 years old) attending upper gastrointestinal endoscopy.
2. Patients able to read and comprehend English.
3. Patients willing and able to provide informed consent.
4. Patients willing and able to provide a venous blood sample.

Exclusion Criteria:

1. Any individual diagnosed with gastric cancer, or with a history of gastric cancer, prior gastrectomy or bariatric surgery.
2. Any individual with a chronic inflammatory condition of the gastrointestinal tract (Crohn's disease or ulcerative colitis).
3. Once enrolment ceiling is reached for each group, enrolment will close for that group. The study will continue until all groups are complete.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for endoscopy within the endoscopy service at participating sites will be invited to participate in the study and provide a blood sample.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-04 (Estimated); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Serologic concentrations of ghrelin, gastrin, pepsinogens and vitamin B12 | Measurements will be made on conclusion of the study, one year after enrollment begins
  Serologic concentrations for patients with atrophic gastritis and intestinal metaplasia will be compared to normal/mild gastritis controls.

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Murphy, PhD MPH, Principal Investigator — Imperial College Dublin

IPD SHARING:
Plan to Share IPD: No